CLINICAL TRIAL: NCT03970668
Title: Linagliptin Plus Insulin for Hyperglycemia Immediately After Renal Transplantation: A Comparative Study
Brief Title: Linagliptin in Post-renal Transplantation
Status: Completed | Type: Observational
Sponsor: Universidad de Guanajuato (Other)
Collaborators: Hospital Regional de Alta Especialidad del Bajio (Other)
Responsible Party: Principal Investigator, Rodolfo Guardado Mendoza, Principal Investigator, Universidad de Guanajuato
Other Study IDs: CEI-49-18
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Transplanted Kidney Complication
MeSH Terms: interventions — Linagliptin; Insulin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Linagliptin plus insulin: Patients that presented hyperglycemia immediately after renal transplantation and received treatment with linagliptin plus insulin
  Interventions: Drug: Linagliptin 5 mg Oral Tablet
- Insulin: Patients that presented hyperglycemia immediately after renal transplantation and received treatment only with insulin
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Linagliptin 5 mg Oral Tablet — Patients received linagliptin 5mg once daily orally plus a basal bolus insulin scheme, if they presented hyperglycemia (glucose levels above than 140 mg/dl)
  Other Names: Linagliptin 5mg once daily plus insulin scheme
  Groups: Linagliptin plus insulin
Drug: Insulin — Patients received a basal bolus insulin scheme, if they presented hyperglycemia (glucose levels above than 140 mg/dl)
  Other Names: Basal bolus insulin scheme
  Groups: Insulin

SUMMARY:
Post-renal transplanted patients frequently present hyperglycemia immediately after the procedure.

This was a retrospective comparative study performed in post-renal transplanted patients in a single high speciality center with the goal of compare the effect of linagliptin + insulin in post-renal transplanted patients with hyperglycemia Interventions were linagliptin 5mg daily plus insulin vs insulin alone during 5 days after renal transplantation with hyperglycemia, and the main outcome were glucose levels, insulin dose and severity of hypoglycemia

DETAILED DESCRIPTION:
This was a retrospective comparative study performed in a single center between 2016 and 2018, included the data collected from 28 hospitalized post-renal transplanted patients that presented hyperglycemia (>140 mg/dl or or 7.77 mmol/l) immediately after renal transplantation (RT); 14 patients were treated with linagliptin 5mg daily plus a basal bolus insulin scheme prescribed by the Endocrinology group at the hospital, and 14 patients treated only with basal bolus insulin scheme were randomly selected from a list of patients treated during the same period of time and by the same Endocrinology group. Linagliptin dose was 5mg daily and the basal bolus insulin regimen was started and adjusted according to the international guidelines; in general, patients received a starting insulin dose of around 0.5 U/kg/day, given half as basal insulin (NPH or Glargine) once or twice daily and half as insulin lispro divided into three equal doses before meals. Insulin dose was adjusted daily to achieve the goal of fasting glucose between 80-140 mg/dl (4.44-7.77 mmol/l) or random glucose levels below 180 mg/dl (9.99 mmol/l). Correctional insulin dose was used before each meal, depending on the glucose measurements, starting at 1 unit for each 40mg above 140 mg/dl (7.77 mmol/l) of glucose. Glucose levels were monitored at fasting and before each meal, as well as at bedtime according to standard clinical practice. Data regarding fasting and preprandial glucose levels, hypoglycemia, renal function, and immunosuppression therapy were recorded from the patient´s file during the first 5 days after RT; fasting glucose and renal function were also recorded at 1, 6 and 12 months after RT. Patients were included if they were between 18-65 years of age and presented fasting hyperglycemia (>140 mg/dl or 7.77 mmol/l) immediately after RT.

Ethical and Research committee (CEI) at the Hospital approved the study protocol with the number CEI-49-18.

ELIGIBILITY:
Inclusion Criteria:

* Hyperglycemia (glucose levels above 140 mg/dl) immediately after renal transplantation

Exclusion Criteria:

* Incomplete records on the patients file
* Acute complications such as liver failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post-transplanted renal patients with hyperglycemia in the hospital setting
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Fasting glucose | 5 days
  Fasting glucose levels at day 5

CONTACTS AND LOCATIONS:
Overall Officials: Rodolfo Guardado, MD, Principal Investigator — Hospital Regional de Alta Especialidad del Bajio

IPD SHARING:
Plan to Share IPD: Undecided
On a specific request we would be able to share data with other researchers

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-30): https://cdn.clinicaltrials.gov/large-docs/68/NCT03970668/Prot_SAP_000.pdf